CLINICAL TRIAL: NCT01320176
Title: An Open-label, Phase I, Dose-escalation and Safety Study of Two Intramuscular Injections of a Dose of 2.9 Log or 4 Log CCID50 of the Recombinant HIV I Clade B Measles Vaccine Vector in Healthy Adults.
Brief Title: Study to Evaluate the Dosage and Safety of Two Intramuscular Injections of an Investigational Clade B HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MV1-F4-CT1
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: HIV

ARMS (2):
- Group A (Experimental): Subjects received dose A of the investigational HIV vaccine
  Interventions: Biological: Investigational HIV vaccine dose A
- Group B (Experimental): Subjects received dose B of the investigational HIV vaccine
  Interventions: Biological: Investigational HIV vaccine dose B

INTERVENTIONS:
Biological: Investigational HIV vaccine dose A — The vaccine will be administered by intramuscular route into the deltoid muscle preferentially of the non dominant arm at Month 0 and Month 3
  Arms: Group A
Biological: Investigational HIV vaccine dose B — The vaccine will be administered by intramuscular route into the deltoid muscle preferentially of the non dominant arm at Month 0 and Month 3
  Arms: Group B

SUMMARY:
This study aimed to evaluate the safety and reactogenicity of two intramuscular injections of two different dosages of an investigational clade B HIV vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) and are available for all scheduled visits at the investigational site
2. Adult male and or female subjects between 18 and 27 years old.
3. Proven record of measles vaccination (longer than 5 years)
4. Measles antibodies titre < 350 IU/L or > 750 IU/L measured in the previous study "CEVAC sero-MV-001".
5. Healthy subjects as established by medical history and clinical examination before entering into the study.
6. Confirmed HIV negative based on the absence of antibodies and p24.
7. Negative for Hepatitis B surface (HBs) antigen, anti-hepatitis B core (HBc antibodies) antibody and anti-Hepatitis C Virus (HCV) antibody

Exclusion Criteria:

1. Participation in another clinical study in the last 6 months in which the subject has been exposed to an investigational product (pharmaceutical product or placebo or device) or concurrent participation in another clinical study during the study period.
2. Previous inclusion in an HIV vaccine study.
3. Receipt of any other vaccination 1 month before or planning to receive any vaccination 1 month after each study vaccination
4. Receipt of tuberculin skin test 1 month before or planning to receive a tuberculin test 1 month after each study vaccination
5. Receipt of allergy treatment with antigen injections 1 month before or planning to receive allergy treatment with antigen injections 1 month after each study vaccination
6. Receipt of blood products or immunoglobulins within 120 days prior to enrolment.
7. Measles vaccination or booster within the last 5 years as confirmed by medical history.
8. Subject is pregnant or breastfeeding or intends to become pregnant within 9 months of enrolling into the study.
9. Subject is of childbearing potential and does not agree to use a medically acceptable form of contraception for the duration of the study (9 months post the first investigational HIV vaccination). Medically acceptable forms of contraception include: Contraceptive Medication, Intrauterine device, Double barrier method (Condom* and Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

   * A female condom and a male condom should not be used together as friction between the two can result in either product failing.
10. History of any significant immunodeficient condition.
11. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the first vaccination
12. Individuals who are at high risk of acquired HIV infection as determined by the risk assessment questionnaire.
13. Individuals who are living and/or working with severely immunocompromised people, children under 15 months old or pregnant women.
14. Family history of immunodeficiency and/or personal history of autoimmune disease (including psoriasis, rheumatoid arthritis, autoimmune thyroid disease).
15. History of type I or type II diabetes mellitus including cases controlled with diet alone.
16. History or ongoing malignancy.
17. Major congenital defects or serious chronic illness at the time of enrolment.
18. History of serious adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the vaccine.
19. Acute or chronic, clinically significant, as determined by the investigator, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
20. Individuals whose Body Mass index (BMI) is less than 18.5 or greater than 30 (i.e. underweight or obese).
21. History of clinically significant, as determined by the investigator, neurological disorder or seizures.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general adverse events (AEs) except fever | 14-day follow-up after each vaccination
Occurrence, intensity and relationship to vaccination of fever | 21-day follow-up after each vaccination
Occurrence, intensity and relationship to vaccination of unsolicited adverse events (AEs) | 42-day follow-up after each vaccination
Occurrence and relationship to vaccination of any serious AEs (SAEs) | During the study period (Month 0-11)
Occurrence, intensity and relationship to vaccination of clinically significant abnormal haematology and biochemistry values (grade 3 or 4) | During the study period (Month 0-11)

SECONDARY OUTCOMES:
Occurrence of shedding of recombinant virus | During the study period (Month 0-11)
Recombinant virus infectivity | During the study period (Month 0-11)
Cell-mediated immune response (CMI) | At day 0, 7, 14, 28, 91, 98, 112, 266
Humoral immune response to HIV antigens | At day 14, 28, 84, 98, 112, 266.

CONTACTS AND LOCATIONS:
Overall Officials: Geert - Leroux-Roels, MD, Principal Investigator — Geert.lerouxRoels@UGent.be
Locations (1):
- Gent University & Hospital, Center for Vaccinology, Ghent, Belgium